CLINICAL TRIAL: NCT03955848
Title: INFUSION OF ALLOREACTIVE NK CELLS AS CONSOLIDATION STRATEGY FOR ADULT ACUTE MYELOID LEUKEMIA PATIENTS: A MULTICENTER CLINICAL STUDY
Brief Title: INFUSION OF ALLOREACTIVE NATURAL KILLER (NK) CELLS AS CONSOLIDATION STRATEGY FOR ACUTE MYELOID LEUKEMIA PATIENTS
Acronym: NKAML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Antonio Curti, Medical Doctor, Hematologist, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35/2017/O/Sper
Record Dates: First submitted 2019-04-12; First posted 2019-05-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Adult Acute Myeloid Leukemia in Remission
Keywords: AML in Remission; NK cells; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM 1 (Experimental): NK cell infusion
  Interventions: Biological: Alloreactive NK cell infusion
- ARM 2 (No Intervention): Follow up without treatment

INTERVENTIONS:
Biological: Alloreactive NK cell infusion — Alloreactive NK cell infusion
  Other Names: Alloreactive NK cells
  Arms: ARM 1

SUMMARY:
Acute Myeloid Leukemia (AML) patients who had achieved Complete Remission (CR) after (re)induction/consolidation chemotherapy will receive the infusion of alloreactive NK cells. Adult AML patients in morphologic, but not cytogenetic and/or molecular CR and AML patients in morphologic plus cytogenetic and/or molecular CR, not eligible for Stem Cell Transplantation (SCT), will be included. Using a genetic randomization through a 'donor' vs 'no donor' approach, patients will undergo NK cell infusion (ARM 1) or followed-up without treatment (ARM 2). Donor alloreactive NK cell repertoire will be evaluated in order to determine the functional cell dose to be used for NK cell collection. NK cells will be selected from a steady-state large volume leukapheresis product from a suitable KIR-ligand incompatible donor. NK cell purification will be performed if the donor leukapheresis product contains at least 10x106 NK cells/Kg, otherwise the final decision for proceeding to NK purification will be made by the PI after careful evaluation of the number of alloreactive If the minimum collected cell dose of 2x105 total alloreactive NK cells/kg is not reached after a single leukapheresis, donors could undergo a second PB collection within 30 days from the first one. Patients will receive immunosuppressive chemotherapy, fludarabine (Flu) 25 mg/mq/ from day -7 to -3 and cyclophosphamide (Cy) 4 g/mq on day -2 (Flu/Cy). Immunosuppressive chemotherapy is not part of the procedures under study and it is used to favor NK cell engraftment. Two days after Cy administration, patients will be infused intravenously with a single dose of cryopreserved NK cells (day 0), which will be followed by subcutaneous administration of Interleuki (IL)-2 (10 x 106 IU/day, 3 times weekly) for 2 weeks (6 doses total). IL-2 administration is not part of the procedures under study and it is used to favor early in vivo expansion of infused NK cells. Peripheral blood samples will be collected for molecular assessment of microchimerism and tracking of NK cells for 30 days, immunophenotype studies, alloreactive NK cells cloning and functional assays. Bone marrow aspirate will be performed once a week until hematological recovery. Enrolled patients (ARM1 and 2) will be followed up for at least 12 months after NK cell infusion. RFS is defined as the time from patient enrollment to disease relapse.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.

  * AML patients in morphologic, but not cytogenetic or molecular CR
  * AML patients in morphologic plus cytogenetic or molecular CR
* Performance Status ≥ 70% (Karnofsky score) or ≤ 2 (WHO)
* Age ≥ 18 years
* Adequate renal (serum creatinine < 2 mg/dl), pulmonary (Sat O2 ≥ 96%) and hepatic function.
* Left Ventricular Ejection Fraction (LVEF) of ≥ 50% as determined by - Echocardiogram

Exclusion Criteria:

* Eligibility to SCT
* Low-risk AML patients in molecular CR
* HIV positivity.
* Hepatiti C Virus positivity (serology and viremia)
* Pregnant or nursing females
* Current uncontrolled infection
* Signs or symptoms of fluid retention (e.g. pleural effusion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2022-05-11 (Estimated)

PRIMARY OUTCOMES:
relapse free survival | 36 months
  relapse-free survival (RFS) of AML patients, not eligible for SCT, who undergo alloreactive NK cell infusion after the achievement of CR with induction/consolidation chemotherapy.
overall survival | 36 months
  overall survival (RFS) of AML patients, not eligible for SCT, who undergo alloreactive NK cell infusion after the achievement of CR with induction/consolidation chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curti, Principal Investigator — Istituto di Ematologia Seràgnoli, Ospedale S.Orsola-Malpighi, Bologna
Locations (1):
- Antonio Curti, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No